CLINICAL TRIAL: NCT07159932
Title: Poland Integrated Medicines Management (PL-IMM) - Randomized Controlled Trial Assessing the Provision of Complex Clinical Pharmacy Services to Hospitalized Patients in the Polish Healthcare System
Brief Title: Poland Integrated Medicines Management (PL-IMM) - Study Assessing the Provision of Complex Clinical Pharmacy Services to Hospitalized Patients
Acronym: PL-IMM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw Medical University (Other)
Responsible Party: Principal Investigator, Kamila Urbańczyk, MPharm, Wroclaw Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KB 47O/2O23N
Record Dates: First submitted 2025-06-24; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Acute Admitted Multimorbid Patients
Keywords: clinical pharmacy; integrated medicines managment; pharmacist interventions; clinical pharmacy services; medicines management; transfer of care; medicines review; medicines reconcilliation; patient education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard care during hospital stay, without pharmacist involved
- Pharmacist intervention - IMM (Experimental): A pharmacist is included in the multidisciplinary treatment team during the hospital stay
  Interventions: Behavioral: multidisciplinary treatment

INTERVENTIONS:
Behavioral: multidisciplinary treatment — The pharmacist will conduct medication reconciliation at admission, perform medication reviews during the hospital stay and provide drug education to the patient before discharge, as well as written drug information
  Arms: Pharmacist intervention - IMM

SUMMARY:
The aim of the study is to assess whether the involvement of a clinical pharmacist in patient care at every stage of hospitalization, from admission to discharge, will improve the quality of healthcare services provided in clinical and economic terms. As part of the research study, we will randomly assign you to two different groups.

Within one group, a pharmacist will be involved in the process of caring for you throughout your hospital stay. The pharmacist will participate in medical rounds, verify medications upon admission to the hospital, check current test results and medical orders regarding pharmacotherapy, verify medications upon discharge and provide advice on the use of medications. All activities will be carried out in consultation with other medical staff. The aim is to check whether such a model of patient care increases safety and leads to improved pharmacotherapy for patients, and also has a positive effect on patient satisfaction and compliance with therapeutic recommendations. Additionally, the opinion of the medical staff and the economic aspects of this solution will be assessed. Within the second group, you will receive standard care offered by the hospital. In the case of both groups, after the hospitalization is completed, the pharmacist will contact you after 1, 3, 6 months to verify your health condition - he or she will ask about any hospitalizations, complications, side effects, and additional visits to the doctor.

DETAILED DESCRIPTION:
Despite the benefits of clinical pharmacy services demonstrated in numerous publications and their implementation in many countries around the world, Poland has still not achieved nationwide implementation. There is also a lack of scientific data at the national level showing the benefits of including a pharmacist in the patient facing activities. Therefore, this RCT aimes to determine if pharmacist input at each stage of hospitalization, from admission to discharge, can result in an enhanced level of patient care when compared to standard care as measured by a number of clinical and economic outcomes. Given the aforementioned, the objective of this research is to:

1. Primary outcome: Determine the incidence of hospital, emergency department and other unscheduled visits after discharge from hospital during the 6 months follow-up period.
2. Secondary outcome: Assess the length of stay (LoS) in hospital.
3. Additional outcomes:

   * Evaluate the service by determining the frequency and type of interventions performed, their acceptance and influence on the quality of pharmacotherapy.
   * Assess the perception of the service by patients.
   * Assess the perception of the service by healthcare professionals.
   * Estimate the potential financial benefits of the service.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting the following inclusion criteria:

• ≥18 years old and an acute admission to the hospital fulfilling at least one of the following criteria:

* taking ≥4 medicines
* taking high risk medicines listed in the medicines reconciliation standard of Polish Society of Clinical Pharmacy (….)
* medicine related admission to the hospital within last 12 months
* chronic kidney or liver disease
* after solid organ transplantation

Exclusion Criteria:

* age below 18 years old
* pregnancy
* resident of long-term care facility
* unable to express informed consent to participate in the research
* expected survival less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Additional episodes of care | 1, 3 and 6 months after discharge
  incidence of hospital, emergency department and other unscheduled visits after discharge from hospital during the 6 months follow-up period

SECONDARY OUTCOMES:
LoS | Periprocedural
  the length of stay (LoS) in hospital

OTHER OUTCOMES:
Interventions | Periprocedural
  Evaluation of the service by determining the type of interventions performed based on classification of French Society of Clinical Pharmacy
Economy | from first patient enrollment at hospital admission until the end of 6 month follow-up period of the last patient enrolled
  Estimation of the potential financial benefits of the service
Patient opinion | at hospital discharge before patient begins the 6 month follow-up period
  The perception of the service by patients based on PSPSQ 2.0 questionnaire
Healthcare team opinion | during the patient's 6 month follow-up period
  The perception of the service by healthcare professionals based on questionnaire prepared by research team
Quality of pharmacotherapy | Periprocedural
  Assessment of quality of pharmacotherapy using PC-MAI

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital in Wroclaw, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided